CLINICAL TRIAL: NCT07397182
Title: SleepSMART for Veterans With Insomnia and Mild Cognitive Impairment: A Randomized Clinical Trial
Brief Title: SleepSMART for Veterans With Insomnia and Mild Cognitive Impairment
Acronym: SleepSMART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RRD4-013-25M; 1I01RD000596-01A2 (Other Grant/Funding Number: VA RRDT)
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Insomnia; Mild Cognitive Impairment
Keywords: Veterans; Insomnia; Mild Cognitive Impairment; Sleep treatment; Cognitive functioning
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two treatment conditions (SleepSMART or CBT-I).
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to treatment condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SleepSMART (Experimental): SleepSMART was developed as an adapted form of CBT-I specifically designed for older Veterans with insomnia and cognitive impairments. SleepSMART focuses on enhancing CBT-I by providing supportive cognitive strategies to boost treatment learning and adherence.
  Interventions: Behavioral: SleepSMART
- CBT-I (Active Comparator): Cognitive Behavioral Therapy for Insomnia (CBT-I) is a structured, evidence-based treatment designed to help individuals overcome chronic insomnia by addressing the underlying cognitive and behavioral factors contributing to sleep difficulties.
  Interventions: Behavioral: Cognitive BehavioralTherapy for Insomnia (CBT-I)

INTERVENTIONS:
Behavioral: Cognitive BehavioralTherapy for Insomnia (CBT-I) — This manualized approach to treatment involves 6 weekly sessions and addresses the underlying causes of insomnia utilizing sleep restriction and stimulus control techniques, relaxation training, and relapse prevention. In Session 1 sleep education, goal setting, and Sleep Restriction Therapy (SRT) guidelines will be introduced. In Session 2 the Veteran's sleep diary will be reviewed, time in bed (TIB) will be modified based on SRT, and Stimulus Control (SC) instructions will be provided. Session 3 will commence with a review of the sleep diary and adjustments to TIB will be made. In this session a discussion of cognitive factors that may impact insomnia and therapy adherence will be discussed. Additionally, stress management and/or relaxation training will be introduced. In Sessions 4 and 5 sleep diaries will be reviewed, adherence to the treatment discussed, and TIB will be modified based on SRT rules. In Session 6 continued care and relapse prevention plans will be developed.
  Arms: CBT-I
Behavioral: SleepSMART — This treatment involves six 50-minute sessions and addresses key CBT-I components including sleep education, sleep restriction/sleep compression therapy, stimulus control techniques, cognitive therapy, relaxation training, and relapse prevention. Each session includes CogSMART cognitive strategies designed to support treatment learning and adherence.
  Arms: SleepSMART

SUMMARY:
Insomnia is a transdiagnostic health problem affecting the physical, cognitive, emotional, and social functioning of Veterans. Importantly, chronic insomnia may be a modifiable risk factor for progression to serious health conditions, such as mild cognitive impairment (MCI) and dementia. Sleep Symptom Management and Rehabilitation Therapy (SleepSMART) was developed as an adapted form of Cognitive Behavioral Therapy for Insomnia (CBT-I) specifically designed for older Veterans with cognitive impairments. SleepSMART focuses on enhancing CBT-I by providing supportive cognitive strategies to boost treatment learning and adherence. In a recent pilot investigation, SleepSMART was found to be feasible, acceptable, and demonstrated preliminary efficacy among a sample of Veterans with co-morbid insomnia and MCI. This proposed investigation aims to conduct a randomized controlled trial investigating the effectiveness of SleepSMART, compared to standard CBT-I in older Veterans with insomnia and MCI.

DETAILED DESCRIPTION:
With increasing age, adults report greater frequency of insomnia symptoms, including difficulty falling and staying asleep, waking too early, and associated impairments in daytime functioning and quality of life. Veterans are particularly vulnerable to insomnia, with rates double and even triple those of civilian populations. When left untreated, chronic insomnia may contribute to increased risk for cognitive decline (e.g., Alzheimer's disease) and can lead to poorer physical health, disruption in major social and occupational responsibilities, and decreased quality of life. CBT-I is the first-line treatment for insomnia, but factors like poor adherence and poor recall for CBT-I content can diminish its impact for certain populations. Specifically, the cognitive impairments experienced by individuals with Mild Cognitive Impairment (MCI) may limit the adherence and rate of progress in CBT-I. Therefore, it is critical to ensure that vulnerable populations, such as older Veterans with MCI, can fully benefit from sleep treatment. The study team developed SleepSMART (Sleep Symptom Management and Rehabilitation Therapy) to help cognitively impaired Veterans learn and adhere to the CBT-I regimen, thereby leading to faster and more complete sleep treatment benefits. Based on the results of a recent pilot investigation, SleepSMART demonstrated preliminary efficacy as a modified form of CBT-I treatment that is uniquely tailored to aging Veterans with MCI. This investigation will build on previous research by conducting a randomized controlled trial investigating the effectiveness of SleepSMART, compared to standard CBT-I, in 150 Veterans age 60+ with insomnia and MCI.

ELIGIBILITY:
Inclusion Criteria:

* Veterans
* chart diagnosis MCI
* DSM-5 diagnosis of insomnia and an Insomnia Severity Index (ISI) score >7 at baseline
* ability to understand, speak, and read English with acceptable visual and auditory acuity
* stable on medications for at least 4 weeks prior to enrollment

Exclusion Criteria:

* presence of neurological disorders such as Parkinson's disease or seizures, dementia (based on chart diagnosis or clear evidence of dementia at the baseline neuropsychological testing using DSM5 criteria for Major Neurocognitive Disorder)
* and/or history of moderate to severe TBI (determined by medical record or self-report of >30 minutes loss of consciousness)
* schizophrenia, psychotic disorder, and/or bipolar disorder
* untreated or poorly managed medical conditions that may impact sleep, including thyroid disease, nocturia, chronic respiratory or heart disease, or diabetes
* untreated obstructive sleep apnea and/or sleep disturbances other than insomnia
* current substance use disorder with <30 days abstinence
* suicidality greater than mild risk as measured by the Columbia-Suicide Severity Rating Scale
* exposure to therapist directed (individual or group) CBT-I within the past year

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2029-11-01 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Pre-treatment (week 1), post-treatment (week 8), and 3-month follow up (week 20)
  Pre-treatment (week 1), post-treatment (week 8), and 3-month follow up (week 20) scores on the ISI will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Almklov, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No